CLINICAL TRIAL: NCT00917072
Title: Innovative Strategies Which Improve the Clinical Handoff (I-SWITCH) Phase II: Randomized Controlled Trial Evaluating Educational Modalities Including Cognitive Simulation
Brief Title: Innovative Strategies Which Improve the Clinical Handoff (I-SWITCH)
Acronym: I-SWITCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Peter Watson, Principle Investigator, Henry Ford Health System
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: HFH-4694
Record Dates: First submitted 2009-06-09; First posted 2009-06-10 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Healthy
Keywords: Clinical Handoff; Medical Education; Simulation; Residency and Internship

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Didactic (Experimental): Group #1: will have a focused, interactive power point lecture on the background, content and guidelines for a good handoff (focus on a standardized electronic hand-off tool). They will have an exercise to complete
  Interventions: Behavioral: Didactic
- Didactic+Simulation (Experimental): Group #2: will undergo the same power point lecture ( as in Group #1) with an additional intervention focused not only on the hand-off tool, but on a standardized hand-off process using an OSCE exercise (objective structured clinical exam). This group will be trained about the effective implementation of the hand-off tool. They will be taught how to standardize the hand-off process and will be given an opportunity to practice with their peers in the HFH simulation center.
  Interventions: Behavioral: Didactic+Simulation
- Control (Placebo Comparator): The control group received no formal handoff training other than an introduction to handoffs for all interns during orientation at the start of the academic year along with expected ward based experiential training from senior residents throughout the intern year.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Didactic — Group #1: will have a focused, interactive power point lecture on the background, content and guidelines for a good handoff (focus on a standardized electronic hand-off tool). They will have an exercise to complete
  Arms: Didactic
Behavioral: Didactic+Simulation — Group #2: will undergo the same power point lecture ( as in Group #1) with an additional intervention focused not only on the hand-off tool, but on a standardized hand-off process using an OSCE exercise (objective structured clinical exam). This group will be trained about the effective implementation of the hand-off tool. They will be taught how to standardize the hand-off process and will be given an opportunity to practice with their peers in the HFH simulation center
  Arms: Didactic+Simulation
Behavioral: Control — The control group received no formal handoff training other than an introduction to handoffs for all interns during orientation at the start of the academic year along with expected ward based experiential training from senior residents throughout the intern year.
  Arms: Control

SUMMARY:
Study the feasibility of different educational modalities to improve resident handoff of patient information b) Determine whether different educational modalities (powerpoint vs. simulation workshop) lead to improved educational and (surrogate) clinical outcomes

1. Educate residents on the content and process of quality handoffs (Medical Knowledge)
2. Educate residents on good communication skills (Communication competency)
3. Improve perceived continuity of patient care, decrease adverse events related to transfer of care. (Patient safety competency)
4. Increase providers (night residents) satisfaction with the continuity of care during handoffs. (system-based practice/ Practice-based learning)

DETAILED DESCRIPTION:
Randomize interns into three groups. The control group has been described above. Two more groups will randomized to one of two interventions: Intervention Group #1: will have a focused, interactive power point lecture on the background, content and guidelines for a good handoff (focus on a standardized electronic hand-off tool). They will have an exercise to complete. Intervention Group #2: will undergo the same power point lecture ( as in Group #1) with an additional intervention focused not only on the hand-off tool, but on a standardized hand-off process using an OSCE exercise (objective structured clinical exam). This group will be trained about the effective implementation of the hand-off tool. They will be taught how to standardize the hand-off process and will be given an opportunity to practice with their peers in the HFH simulation center. Up to 12 residents will be taken in pairs to practice written and verbal handoff skills in the simulation center under peer observation and by faculty (investigators, PI). Each intern will be given a simulated patient history and physical and any relevant information related to the patient's hospital course. The intern will be given five minutes to create a handoff. Each pair will go into a separate room that will be recorded and viewed by their peers and instructor. They will be observed giving a handoff and receiving a handoff. When they exit the room, they will provide feedback to one another regarding the quality of the handoff. Then the peers will give additional feedback. Each intern will go through the process of giving a handoff and the one accepting the handoff. After the simulation, they will complete a short survey on the intervention. At the completion of the educational interventions, throughout the year as part of regular intern evaluations, night residents will be asked on a weekly basis to evaluate the efficacy of intern handoffs. In addition, de-identified written handoffs will be evaluated by the investigators and scored for completeness and accuracy. The resident cross covering will be blinded to the intern group. They will evaluate the handoff process. During this process, content omission can be measured, as well as time taken to cross cover a patient.

All interns participating in the study will do a self-assessment of their handoff skills. Interns will then be randomized into one of three groups as described above and undergo the educational intervention (#1 or #2) or standard education (control). Educational interventions will be completed within 10 days of the start of the study (Specific Aims #1,2). Following the interventions interns will be assessed throughout the year using a standardized grading form that evaluates written and verbal handoff skills, and perceived effectiveness of handofffs and it pertains to patient care for interns on inpatient rotations that month (Specific Aim #3,4). This will be completed on a weekly basis by night residents (second and third year residents not involved in the study, and blinded to the intervention groups). Educational endpoints: perceived improvement in handoff skills by interns involved in the study over a 6 month period of time as compared among the intervention groups. (Surrogate) Clinical Endpoints: 1) Objective handoff skills evaluation of interns by more senior residents using a standardized grading form 2) Review of electronic handoff forms by investigators, forms by individual interns will be blinded to the investigators to reduce bias

ELIGIBILITY:
Inclusion Criteria:

* Inclusion: interns starting July 1st 2007 in the internal medicine program and including EM/IM residents starting in July 1st, 2007. All residents will participate as part of an ongoing quality improvement project in the internal medicine curriculum.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2007-09; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Critical missed events or 'surprises' overnight due to an inadequate or unclear handoff (errors/intern/night), as determined by nightfloat residents | daily for 3 month study period

SECONDARY OUTCOMES:
nightfloat residents' overall judgment on the handoff quality and observed verbal and written handoff performance by interns | daily, over 3 month study period
interns' knowledge and attitudes on their handoff performance | pre-intervention, and 30 days post-intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

REFERENCES:
- [Result] Han, Jenny; Lukowski, Anna; Watson, Peter. Innovative Strategies Which Improve the Clinical Handoff (I-SWITCH) Phase II: Randomized Controlled Trial Evaluating Educational Modalities Including Cognitive Simulation. The Journal of Hospital Medicine. 2009;4(s1):26